CLINICAL TRIAL: NCT07027605
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Performance Improvement From Computer-aided Tool for the Prognostic Prediction of Colorectal Liver Metastases
Brief Title: Multi-Reader Multi-Case Trial Evaluating Computer-Aided Tool for Prognostic Prediction of Colorectal Liver Metastases
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC-017834
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Liver Metastasis (CRLM)
Keywords: Multi-Reader Multi-Case Controlled Clinical Trial; Prognostic Prediction; Colorectal Liver Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reader Group A: Interprets Dataset A in unaided scenario and Dataset B in aided scenario: A reader study with 12 readers (4 Junior Physician, 4 mid-level Physician and 4 Senior Physician) from the Department of Surgical Oncology of the Digestive Tract will be conducted. The readers are equally and randomly split between Group A and Group B. The study will target 166 CRLM patient cases receiving simultaneous resection.Patient cases will be equally and randomly split between Dataset A and Dataset B.
- Reader Group B: Interprets Dataset A in aided scenario and Dataset B in unaided scenario: A reader study with 12 readers (4 Junior Physician, 4 mid-level Physician and 4 Senior Physician) from the Department of Surgical Oncology of the Digestive Tract will be conducted. The readers are equally and randomly split between Group A and Group B. The study will target 166 CRLM patient cases receiving simultaneous resection.Patient cases will be equally and randomly split between Dataset A and Dataset B.

SUMMARY:
This study evaluates the impact of a novel computer-aided prognostic prediction tool for colorectal liver metastases (CRLM) on clinician performance. Colorectal cancer is a leading cause of cancer-related mortality worldwide, with 20-30% of patients presenting synchronous liver metastases, which are associated with poor prognosis and high postoperative recurrence rates. Simultaneous resection of primary tumor and liver metastases is a preferred treatment for selected patients but outcomes vary significantly. The latest web-based tool uses Random Forest models integrating demographic, clinical, laboratory, and genetic data to predict postoperative recurrence and mortality specifically for CRLM patients undergoing simultaneous resection. This multiple-reader, multiple-case (MRMC) study will assess 12 physicians who will predict 1-, 3-, and 5-year recurrence and mortality risks in 166 retrospective cases, with and without the tool's aid, separated by a washout period. The primary focus is to determine whether the tool improves prediction accuracy for 3-year postoperative mortality, measured by AUC-ROC. Secondary and exploratory endpoints include other time points, sensitivity, specificity, inter-rater reliability, decision-making confidence, and evaluation time. By enabling individualized risk assessment, this tool aims to support optimized clinical decision-making and tailored treatment strategies for CRLM patients undergoing simultaneous resection.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of a novel computer-aided prognostic prediction tool on clinician performance in managing patients with colorectal liver metastases (CRLM). Colorectal cancer remains one of the leading causes of cancer-related mortality worldwide, with approximately 20-30% of patients presenting synchronous liver metastases at diagnosis. These metastases are associated with poor prognosis and a high rate of postoperative recurrence.

For selected patients, simultaneous resection of the primary colorectal tumor and liver metastases is the preferred treatment approach, though clinical outcomes vary widely. To address this variability, the latest web-based prediction tool employs Random Forest machine learning models that integrate comprehensive demographic, clinical, laboratory, and genetic data. This tool is specifically designed to predict postoperative recurrence and mortality for CRLM patients undergoing simultaneous resection, enabling individualized risk assessment.

In this multiple-reader, multiple-case (MRMC) study, 12 physicians will independently evaluate 166 retrospective patient cases. Each physician will estimate the risk of disease recurrence and mortality at 1-, 3-, and 5-year time points, both with and without access to the prediction tool. These two assessment phases will be separated by a washout period to minimize bias.

The primary objective is to determine whether use of the tool improves the accuracy of predicting 3-year postoperative mortality, quantified by the area under the receiver operating characteristic curve (AUC-ROC). Secondary and exploratory endpoints include prediction accuracy at other time points, sensitivity, specificity, inter-rater reliability, clinician confidence in decision-making, and time required for evaluation.

By providing specific, data-driven risk estimates, this computer-aided prognostic tool aims to enhance clinical decision-making and support personalized treatment planning for CRLM patients undergoing simultaneous resection, ultimately striving to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* confirmation of histologically diagnosed liver metastases of colorectal adenocarcinoma
* receiving colorectal resection with simultaneous liver resection.

Exclusion Criteria:

* presence of other malignancies
* absence of follow-up data
* patients who were followed up postoperatively for less than 5 years and had no occurrences of death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This reader study involves 12 physicians (4 junior, 4 mid-level, 4 senior) from the Surgical Oncology Department of the Digestive Tract. All readers will receive standardized training on accessing patient data through the medical record system and completing the questionnaire. The study includes 166 colorectal liver metastases (CRLM) patients who underwent simultaneous colorectal and liver resection. Inclusion criteria: age ≥18 years, histologically confirmed colorectal adenocarcinoma liver metastases, and simultaneous resection. Exclusion criteria: presence of other malignancies, lack of follow-up data, or postoperative follow-up less than 5 years without death occurrence.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
AUCs: Area Under the Receiver Operating Characteristic Curve (AUC-ROC) | Up to approximately 120 months
  The comparative accuracy of model aided versus unaided risk prediction of post-operative 3-year mortality assessed by readers. Under model aided condition, prediction model will estimate the overall survival (OS) rate at Year 3 for each individual patient. OS was defined as the time from the date of simultaneous resection to death due to any cause. Patients without death were censored at their last known alive date. The mortality data were retrospectively collected and the event status were known. Patients were followed up to approximately 120 months after simultaneous resection.

SECONDARY OUTCOMES:
AUCs: Area Under the Receiver Operating Characteristic Curve (AUC-ROC) | Up to approximately 120 months
  The comparative accuracy of model aided versus unaided risk prediction of post-operative 1-year recurrence, 3-year recurrence, 5-year recurrence, 1-year mortality, and 5-year mortality made by readers.
  PFS was defined as the time from the date of simultaneous colorectal and liver resection to first documented disease progression or death due to any cause, whichever occurs first. Patients without PFS event were censored at their last assessment follow-up.
  OS was defined as the time from the date of simultaneous resection to death due to any cause. Patients without death were censored at their last known alive date.
  Patients were followed up to approximately 120 months after simultaneous resection.
Sensitivity: the ratio of true positives to total (actual) positives. | Up to approximately 120 months
  To evaluate aided versus unaided with respect to (improved) sensitivity for prediction of post-operative 1-year, 3-year, and 5-year recurrence and mortality made by readers.
Specificity: the ratio of true negatives to total (actual) negatives. | Up to approximately 120 months
  To evaluate aided versus unaided with respect to (improved) specificity for prediction of post-operative 1-year, 3-year, and 5-year recurrence and mortality made by readers.
Inter-rater reliability: the consistency of ratings made by readers on the cases | Up to approximately 120 months
  To evaluate aided versus unaided with respect to (improved) inter-rater reliability for rating on the likelihood of post-operative 1-year, 3-year, and 5-year recurrence and mortality made by readers.

OTHER OUTCOMES:
Inter-rater reliability: the consistency of ratings made by readers on the cases | Up to approximately 120 months
  To evaluate aided versus unaided with respect to inter-rater reliability for readers' recommendation on initiating surgical treatment; To evaluate aided versus unaided with respect to inter-rater reliability for readers' recommendation on the timing of the first post-surgery follow-up.
Decision-making confidence: confidence of a reader in completing the evaluation for a case | Up to approximately 120 months
  To evaluate aided versus unaided with respect to (improve) decision-making confidence in predicting the disease progression and making recommendation for a case. The general confidence on prediction model in pre and post study will also be evaluated.
Decision-making time: duration of a reader in completing the evaluation for a case | Up to approximately 120 months
  To evaluate aided versus unaided with respect to (reduced) decision-making time in completing a case evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhao, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- No. 17, South Panjiayuan, Chaoyang District, Beijing, Cancer Hospital, Chinese Academy of Medical Sciences, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Imai K, Allard MA, Castro Benitez C, Vibert E, Sa Cunha A, Cherqui D, Castaing D, Bismuth H, Baba H, Adam R. Nomogram for prediction of prognosis in patients with initially unresectable colorectal liver metastases. Br J Surg. 2016 Apr;103(5):590-9. doi: 10.1002/bjs.10073. Epub 2016 Jan 18. PMID 26780341
- [Result] Chen Q, Deng Y, Li Y, Chen J, Zhang R, Yang L, Guo R, Xing B, Ding P, Cai J, Zhao H. Association of preoperative aspartate aminotransferase to platelet ratio index with outcomes and tumour microenvironment among colorectal cancer with liver metastases. Cancer Lett. 2024 Apr 28;588:216778. doi: 10.1016/j.canlet.2024.216778. Epub 2024 Mar 6. PMID 38458593
- [Result] Wu Y, Mao A, Wang H, Fang G, Zhou J, He X, Cai S, Wang L. Association of Simultaneous vs Delayed Resection of Liver Metastasis With Complications and Survival Among Adults With Colorectal Cancer. JAMA Netw Open. 2022 Sep 1;5(9):e2231956. doi: 10.1001/jamanetworkopen.2022.31956. PMID 36121654
- [Result] Kataoka K, Takahashi K, Takeuchi J, Ito K, Beppu N, Ceelen W, Kanemitsu Y, Ajioka Y, Endo I, Hasegawa K, Takahashi K, Ikeda M. Correlation between recurrence-free survival and overall survival after upfront surgery for resected colorectal liver metastases. Br J Surg. 2023 Jun 12;110(7):864-869. doi: 10.1093/bjs/znad127. PMID 37196147
- [Result] Machairas N, Di Martino M, Primavesi F, Underwood P, de Santibanes M, Ntanasis-Stathopoulos I, Urban I, Tsilimigras DI, Siriwardena AK, Frampton AE, Pawlik TM. Simultaneous resection for colorectal cancer with synchronous liver metastases: current state-of-the-art. J Gastrointest Surg. 2024 Apr;28(4):577-586. doi: 10.1016/j.gassur.2024.01.034. Epub 2024 Feb 9. PMID 38583912
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Result] Chen Q, Chen J, Deng Y, Bi X, Zhao J, Zhou J, Huang Z, Cai J, Xing B, Li Y, Li K, Zhao H. Personalized prediction of postoperative complication and survival among Colorectal Liver Metastases Patients Receiving Simultaneous Resection using machine learning approaches: A multi-center study. Cancer Lett. 2024 Jul 1;593:216967. doi: 10.1016/j.canlet.2024.216967. Epub 2024 May 18. PMID 38768679

DOCUMENTS (1):
  • Study Protocol (2025-06-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT07027605/Prot_001.pdf